CLINICAL TRIAL: NCT02701621
Title: Aquatic Therapy Versus Land-Based Therapy for the Treatment of Balance Dysfunction in Parkinson's Disease: a Randomized, Controlled Study With 6-months Follow-up
Brief Title: Aquatic Therapy Versus Land-Based Therapy for the Treatment of Balance Dysfunction in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATvsLB Therapy for BD in PD
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease, aquatic therapy, balance, MIRT
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIRT Group (Active Comparator): Individuals underwent Multidisciplinary Intensive Rehabilitation Treatment. It consists of 4 weeks of physical therapy in a hospital setting with four daily sessions for five days and one hour of physical exercise on the sixth day.The duration of each session is about one hour. The first session comprises cardiovascular warm-up activities, relaxation and muscle-stretching. The second session includes aerobic exercises and the use of different devices: a stabilometric platform, treadmill plus, crossover, cycloergometer. The third is a session of occupational therapy. The last session includes one hour of speech therapy. The rehabilitation program can also include: robotic-assisted walking training, virtual reality training and meetings with a Psychologist.
  Interventions: Other: MIRT
- MIRT-AT (Experimental): Patients underwent land-based therapy in association with aquatic therapy, three times per week for four weeks.
  The land-based activities included the second and the third session of MIRT.
  The water sessions were divided in 3 phases:
  i) Warm Up Exercises. This phase lasted 10 minutes and comprised walking performances.
  ii) Central session Training. This phase lasted 30-45 minutes and comprised trunk mobility exercises in standing position and sitting on a floating device, static and dynamic exercises. The successive balance training exercises comprised: maintaining balance with closed eyes; balance control with one leg resting on a step; postural control changing the support base.
  iii) Cool-down. This phase lasted 5 minutes and comprised general stretching exercises and gentle walking.
  Interventions: Other: MIRT-AT

INTERVENTIONS:
Other: MIRT-AT — Aquatic therapy
  Arms: MIRT-AT
Other: MIRT — Land-based Therapy
  Arms: MIRT Group

SUMMARY:
The aim of this study is to compare the effectiveness of a specific aquatic therapy program on balance with a land-based physical-treatment in patients with Parkinson's disease and to evaluate the long-term effects in a 6-month follow-up period.

DETAILED DESCRIPTION:
Background: Balance dysfunction (BD) in Parkinson's disease (PD) is a disabling sign leading to falls which have a negative impact on the quality of life. It is known that aquatic therapy could be useful to train balance given its physical features and for reducing patients' fear of falls. Many studies have evaluated the efficacy of land-based physiotherapy in treatment of BD, but few studies have investigated the efficacy of aquatic therapy on balance and none of those assessed clinical measurements in a clinically, relevant follow-up period.

Objective: The aim of study was to compare the effectiveness of a specific aquatic therapy program on balance with a land-based physical-treatment in patients with PD and to evaluate the long-term effects in a 6-month follow-up period.

Methods: Thirty-four patients with PD in medium-stage of disease were randomized into two groups: 17 underwent Multidisciplinary-Intensive-Rehabilitation-Treatment (MIRT) and 17 underwent MIRT associated with aquatic therapy protocol (MIRT-AT). Investigators assessed the Berg Balance Scale (BBS), Unified Parkinson's Disease Rating Scale (UPDRS) II-III, and Timed Up Go test (TUG) in both groups at admission, discharge and after a 6-months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Probable diagnosis of PD according to Gelb et al
* Hoehn & Yahr stage 2.5-3 (H&Y),
* Stable pharmacological treatment for the last 8 weeks and during the hospitalization
* Mini-Mental State Examination (MMSE) ≥ 24

Exclusion Criteria:

* Cardiac and pulmonary diseases
* Urinary incontinence
* History of deep brain stimulation

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 6 months

SECONDARY OUTCOMES:
TUG | 6 months
Unified Parkinson's Disease Rating Scale II | 6 months
Unified Parkinson's Disease Rating Scale III | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital - Gravedona ed Uniti (CO, Italy)
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palamara G, Gotti F, Maestri R, Bera R, Gargantini R, Bossio F, Zivi I, Volpe D, Ferrazzoli D, Frazzitta G. Land Plus Aquatic Therapy Versus Land-Based Rehabilitation Alone for the Treatment of Balance Dysfunction in Parkinson Disease: A Randomized Controlled Study With 6-Month Follow-Up. Arch Phys Med Rehabil. 2017 Jun;98(6):1077-1085. doi: 10.1016/j.apmr.2017.01.025. Epub 2017 Feb 27. PMID 28254636